CLINICAL TRIAL: NCT04986072
Title: Proof of Mechanism Study Using a Retinal Biomarker to Predict Treatment Response With Intravenous Sodium Nitroprusside in Symptomatic Early Course Schizophrenia
Brief Title: Sodium Nitroprusside in Early Course Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with recruiting subjects for the study
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Paulo Lizano, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK3831-A309
Record Dates: First submitted 2021-07-23; First posted 2021-08-02 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Nitroprusside; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Nitroprusside Arm (Experimental): Sodium Nitroprusside (0.5 μg/kg/min) for 4 hours
  Interventions: Drug: Sodium Nitroprusside
- Placebo Arm (Placebo Comparator): 5% Dextrose (0.5 μg/kg/min) for 4 hours
  Interventions: Drug: 5% Dextrose solution

INTERVENTIONS:
Drug: Sodium Nitroprusside — Half of participants will receive Intravenous Sodium Nitroprusside (0.5 μg/kg/min) for 4 hours.
  Other Names: Active
  Arms: Sodium Nitroprusside Arm
Drug: 5% Dextrose solution — Half of participants will receive intravenous 5% Dextrose solution for 4 hours.
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
Peripheral inflammation and microvascular dysfunction are central to the pathophysiology of schizophrenia (SZ). Retinal imaging allows for the accurate quantitative assessment of the condition of retinal microvessels, and early studies implicate microvascular dysfunction in SZ, but the specific pathophysiological mechanisms underlying greater length, density, capillary network and diameter are not yet entirely understood. Anti-inflammatory drug trials in SZ suggest that Early Course Schizophrenia (ECS) individuals with elevated peripheral inflammation show the greatest benefit to adjunctive anti inflammatory treatments. Also, there is a growing interest in the use of Sodium Nitroprusside (SNP) in SZ but further studies are needed as results are inconsistent. This study will determine the effectiveness of SNP on psychosis symptoms, cognition, and retinal measures in symptomatic ECS.

DETAILED DESCRIPTION:
The microvascular environment is the major interface of systemic factors affecting the brain, it is a logical focus for understanding the neurobiology of schizophrenia (SZ). However, our understanding of the immunological underpinnings of SZ and improved methodologies to detect microvascular disorder have led to increased research in this area. We have shown that inflammatory subtypes are found in psychosis and an increased pattern of peripheral inflammation (including C-Reactive Protein, CRP) is related with worse overall cognition. Retinal and cerebral microvessels are embryological related and can be utilized to measure the state of cerebral microvessels. Advances in retinal imaging, such as swept source optical coherence tomography angiography (SS-OCTA), provide greater microvascular clarity to visualize the retina non-invasively, in a more detailed, quicker and cost-effective manner. In a pilot study using SS-OCTA, we identified microvascular dysfunction associated with early-stages SZ. The pathophysiological mechanisms underlying these retinal microvascular changes are not entirely understood, but they have been associated with inflammation (including CRP), endothelial dysfunction, reactive oxygen species and hypoxia/ ischemia, which have also been consistently observed in SZ. Nitric oxide (NO) signaling is a potential mechanism for protecting the microvasculature against oxidative stress, inflammation and endothelial dysfunction and treatment with NOD have been shown to reduce oxidative stress/inflammation and to increase cerebral blood flow in cerebrovascular disorders. Anti-inflammatory drug trials in SZ suggest that Early Course Schizophrenia (ECS) individuals with elevated peripheral inflammation show the greatest benefit to adjunctive anti inflammatory treatments. In line with that there is a growing interest in the use of SNP in SZ. Preclinical and clinical evidence have shown that SNP may have an antipsychotic profile. Hallak et al (2013) demonstrated that a single infusion of SNP in patients with ECS was both safe and associated with immediate and longer-term clinical outcome. While three other studies demonstrated that SNP was well-tolerated in patient with multi-episode SZ, they were not able to replicate Hallak's finding, which was likely due to the disease heterogeneity, the inclusion of an older population with a longer duration or multi-episodes of illness, and the lack of treatment biomarkers. Further work is needed to determine whether the effect of SNP treatment is dependent on a patient's illness duration and whether a retinal biomarker for microvascular dysfunction/inflammation can predict treatment response to SNP. Thus, the principal goal in the field of SZ is to identify biomarker-based targets for early intervention, evidence of engaging this target by selective interventions and assessing therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Having a DSM-V diagnosis of Schizophrenia or schizoaffective disorder with <5 years from the onset of psychosis
* Having up to 2 years of lifetime exposure to antipsychotics
* Having total score of >65 on the Positive and Negative Syndrome Scale (PANSS) with a score of >4 on 1 or more PANSS items (delusions, conceptual disorganization, hallucinatory behavior, suspiciousness, or unusual thought content)
* Having English proficiency
* Being competent and willing to give informed consent

Exclusion Criteria:

* Having substance dependence or abuse within the past 6 months
* Having history of retinal disease; myopia >4.0 diopters; symptomatic orthostatic hypotension
* Any change of psychotropic medications within the previous 4 weeks
* Currently taking clozapine
* Having prior history of intolerance to Sodium Nitroprusside
* Having treatment with medications that may interfere with the metabolism or excretion or effects of Sodium Nitroprusside
* Being pregnancy/breast feeding
* Having unstable major medical (renal, hepatic, or cardiac) or neurologic illness
* Having significant inflammatory or immune conditions
* Having treatment with anti-inflammatory drugs, hormones or immunosuppressant agents in the 6 months before study entry.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Lizano, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: study terminated sue to low recruitment
Period: Overall Study
Arm/Group | Sodium Nitroprusside Arm | Placebo Arm
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study Terminated due to low enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Nitroprusside Arm | Placebo Arm | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Customized [Count of Participants; unit: Participants]
  Due to privacy concerns of single participant, data will not be shown for this outcome |  | NA — Due to privacy concerns of single participant, data will not be shown for this outcome | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Due to privacy concerns of single participant, data will not be shown for this outcome |  | NA — Due to privacy concerns of single participant, data will not be shown for this outcome | NA — Total not calculated because data are not available (NA) in one or more arms.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 0 | 0
  Unknown or Not Reported |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1
PANSS Total Score [Number; unit: score on scale] — Due to privacy concerns of single participant, data will not be shown for this outcome.
  score on scale |  | NA — Due to privacy concerns of single participant, data will not be shown for this outcome | 0

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: Comparing total, positive, and negative scores between SNP and Placebo
Time Frame: Measured at hour 2
Population: Due to privacy concerns of single participant, data will not be shown for this outcome
Arm/Group | Sodium Nitroprusside Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collect up to 4 weeks after intervention
Description: Due to low recruitment efforts the study was terminated. Only 1 individual participated and was allocated to the placebo arm.
Arm/Group | Sodium Nitroprusside Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Due to privacy concerns of single participant, data will not be shown for this outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT04986072/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT04986072/ICF_001.pdf